CLINICAL TRIAL: NCT00071981
Title: A Randomized Phase II Trial of Multi-Epitope Vaccination With Melanoma Peptides For Cytotoxic T Cells And Helper T Cells For Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy Using Melanoma Peptides for Cytotoxic T Cells and Helper T Cells in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000335055; U10CA021115 (NIH); E1602 (Other: Eastern Cooperative Oncology Group (ECOG)); NCT00464152 (obsolete NCT alias)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; montanide ISA 51; dipeptidase 1; sargramostim; Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (12MP) (Experimental): Patients receive 2 injections of multi-epitope peptide vaccine comprising 12 melanoma peptides restricted by Class I MHC (12MP) emulsified with sargramostim (GM-CSF) and Montanide ISA-51 (incomplete Freund's adjuvant) or Montanide ISA-51 VG (ISA-51) intradermally (ID) and subcutaneously (SC) on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: multi-epitope melanoma peptide vaccine; Biological: sargramostim
- Arm II (12MP/Tet) (Experimental): Patients receive 2 injections of multi-epitope peptide vaccine comprising multi-epitope melanoma peptide vaccine (12MP) and 1 tetanus peptide melanoma vaccine emulsified with GM-CSF and ISA-51 (incomplete Freund's adjuvant) ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: multi-epitope melanoma peptide vaccine; Biological: sargramostim; Biological: tetanus peptide melanoma vaccine
- Arm III (12MP/6MHP) (Experimental): Patients receive 2 injections of multi-epitope peptide vaccine comprising multi-epitope melanoma peptide vaccine (12MP) and 6 melanoma helper peptides (6HP) emulsified with GM-CSF and ISA-51 (incomplete Freund's adjuvant) ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: melanoma helper peptide vaccine; Biological: multi-epitope melanoma peptide vaccine; Biological: sargramostim
- Arm IV (6MHP) (Experimental): Patients receive 2 injections of multi-epitope peptide vaccine comprising melanoma helper peptide vaccine (6HP) emulsified with GM-CSF and ISA-51 (incomplete Freund's adjuvant) ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: melanoma helper peptide vaccine; Biological: sargramostim

INTERVENTIONS:
Biological: incomplete Freund's adjuvant — Given by injection
  Other Names: Montanide ISA-51
Biological: melanoma helper peptide vaccine — Given by injection
  Other Names: 6 melanoma helper peptides restricted by class II MHC molecules, restricted by; HLADR molecules,; 6 class II MHC-Restricted Melanoma-Associated Peptides
  Arms: Arm III (12MP/6MHP); Arm IV (6MHP)
Biological: multi-epitope melanoma peptide vaccine — Given by injection
  Other Names: 12 Melanoma peptides from melanocyte differentiation protein (MDP) and cancer testis antigen (CTA),; 12 melanoma peptides restricted by class I MHC molecules,restricted by HLA-A1, A2, or A3 molecules
  Arms: Arm I (12MP); Arm II (12MP/Tet); Arm III (12MP/6MHP)
Biological: sargramostim — Given by injection
  Other Names: rhu GM-CSF,; Leukine,; Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF)
Biological: tetanus peptide melanoma vaccine — Given by injection
  Other Names: Modified Tetanus p2 peptide restricted by class II MHC molecules,; Peptide-Tet
  Arms: Arm II (12MP/Tet)

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response to kill tumor cells.

PURPOSE: This randomized phase II trial is studying four different vaccines using melanoma peptides from cytotoxic T cells and helper T cells to see how well they work in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the cytotoxic T-cell response to each of 12 melanoma peptides restricted by Human Leukocyte Antigen (HLA)-A1, -A2, or -A3 in patients with metastatic melanoma vaccinated with or without these 12 melanoma peptides and with or without helper peptides.
* Compare the helper T-cell response to each of 6 melanoma helper peptides restricted by HLA-DR molecules in patients treated with these vaccinations.
* Determine whether the addition of 6 melanoma helper peptides to a vaccine containing multiple class I Major histocompatibility complex (MHC)-restricted peptides augments T-cell responses to the class I restricted peptides in these patients.
* Determine, preliminarily, whether booster vaccination maintains immune response in patients treated with these vaccinations.
* Compare the rates of clinical response and survival in patients treated with these vaccinations.
* Determine, preliminarily, whether cellular immune response correlates with clinical response and survival rates in patients treated with these vaccinations.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to HLA type (HLA-A1 vs HLA-A2 vs HLA-A1 and -A2 vs HLA-A3) and planned sentinel immunized node biopsy (yes vs no). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive 2 injections of multi-epitope peptide vaccine comprising 12 melanoma peptides restricted by Class I MHC (12MP) emulsified with sargramostim (Granulocyte-macrophage colony-stimulating factor, GM-CSF) and Montanide ISA-51 or Montanide ISA-51 VG (ISA-51) intradermally (ID) and subcutaneously (SC) on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
* Arm II: Patients receive 2 injections of multi-epitope peptide vaccine comprising 12MP and 1 tetanus helper peptide emulsified with GM-CSF and ISA-51 ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
* Arm III (closed to accrual as of 5/19/08): Patients receive 2 injections of multi-epitope peptide vaccine comprising 12MP and 6 melanoma helper peptides (6HP) emulsified with GM-CSF and ISA-51 ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
* Arm IV: Patients receive 2 injections of multi-epitope peptide vaccine comprising 6HP emulsified with GM-CSF and ISA-51 ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.

In all arms, patients continue therapy in the absence of unacceptable toxicity or disease progression necessitating other urgent therapy.

Patients are evaluated at 8 and 12 weeks. Beginning 2-3 weeks after the week-12 evaluation, patients with no evidence of disease progression may receive booster vaccinations according to their randomized treatment arm. Patients receive booster vaccination ID and SC once weekly for 3 weeks. Treatment repeats every 9 weeks for 1 course, every 12 weeks for 2 courses, and then every 24 weeks for 2 courses OR for up to 2 years (whichever comes first) provided the patient does not require an urgent change in therapy.

After completion of study treatment, patients are followed every 6 months for 2 years and then for survival for 5 years from study randomization.

ACTUAL ACCRUAL: A total of 175 patients were accrued for this study during March 2005 and January 2009.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV melanoma

  * Multiple primary melanomas allowed
  * Metastasis may be from a cutaneous, mucosal, ocular, or unknown primary site
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST criteria)
* Must have 2 extremities uninvolved with tumor
* Must have at least 2 intact (undissected) axillary and/or inguinal lymph node basins

  * Prior sentinel node biopsy may not have violated the integrity of a nodal basin

    * This extremity may still be considered for vaccination
* Human Lymphocyte Antigen (HLA)-A1, -A2, or -A3 positive
* Prior brain metastases allowed provided all of the following are true:

  * Surgically resected or treated with gamma-knife or stereotactic radiosurgery
  * No disease progression in the brain for the past 3 months
  * More than 30 days since prior steroids for the management of brain metastases
* Age: 18 and over
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate organ function measured within 4 weeks before randomization:

  * White blood cell (WBC) at least 4,000/mm^3
  * Platelet count at least 100,000/mm^3
  * Lymphocyte count at least 700/mm^3
  * Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) no greater than 2 times upper limit of normal (ULN)
  * Bilirubin no greater than 2 times ULN
  * Alkaline phosphatase no greater than 2 times ULN
  * Lactic dehydrogenase no greater than 2 times ULN
  * Creatinine no greater than 1.8 mg/dL
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmetastatic squamous cell or basal cell skin cancer, ductal or lobular carcinoma in situ of the breast, or carcinoma in situ of the cervix
* At least 4 weeks since prior sargramostim (GM-CSF), interferon alfa-2b, or interleukin-2
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 30 days since prior systemic corticosteroids, including any of the following:

  * Therapeutic doses of oral steroids (e.g., prednisone or dexamethasone)
  * Steroid inhalers (e.g., Advair)

    * Topical steroids and nasal steroids with low systemic absorption (e.g., fluticasone) or steroids with low systemic absorption (e.g., triamcinolone hexacetonide) injected into a joint space allowed
* At least 4 weeks since prior local control or palliative radiotherapy and recovered
* Recovered from prior major surgery

Exclusion criteria:

* More than 3 brain metastases
* Metastatic lesions greater than 2 cm
* Concurrent radiotherapy
* Prior radiotherapy to measurable disease
* Concurrent surgery
* Concurrent corticosteroids
* Concurrent topical or systemic steroids
* Concurrent chemotherapy
* Prior vaccination with any of the study peptides
* Recent (within the past year) or concurrent addiction to alcohol or illicit drugs
* Pregnant or nursing
* Known or suspected major allergy to any components of the study vaccine
* Significant detectable infection
* Immunosuppression conditions
* Prior or active autoimmune disorder requiring cytotoxic or mmunosuppressive therapy, except for any of the following:

  * Presence of laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody (ANA) titer) without symptoms
  * Clinical evidence of vitiligo or other forms of depigmenting illness
  * Mild arthritis requiring nonsteroidal anti-inflammatory medication
* Autoimmune disorder with visceral involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2005-05-09 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Study Chair — University of Virginia
Locations (65):
- United States (65):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford Cancer Center, Stanford, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on March 21, 2005, accrued its first patient on May 9, 2005, and terminated on January 12, 2009 with the final accrual of 175 patients.22 ECOG institutions participated in the study.
Pre-assignment Details: This study involved a pre-registration before randomization. For patients with locally-typed HLA status, randomization immediately followed pre-registration. For central evaluation of HLA status, samples were submitted after pre-registration, and results of the evaluation must have been received from the central laboratory prior to randomization
Groups:
- Arm I (12MP): Patients receive 2 injections of multi-epitope peptide vaccine comprising 12 melanoma peptides restricted by Class I MHC (12MP) emulsified with sargramostim (GM-CSF) and Montanide ISA-51 (incomplete Freund's adjuvant) or Montanide ISA-51 VG (ISA-51) intradermally (ID) and subcutaneously (SC) on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  multi-epitope melanoma peptide vaccine : Given by injection
  incomplete Freund's adjuvant : Given by injection
  sargramostim : Given by injection
- Arm II (12MP/Tet): Patients receive 2 injections of multi-epitope peptide vaccine comprising multi-epitope melanoma peptide vaccine (12MP) and 1 tetanus peptide melanoma vaccine emulsified with GM-CSF and ISA-51 (incomplete Freund's adjuvant) ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  multi-epitope melanoma peptide vaccine : Given by injection
  incomplete Freund's adjuvant : Given by injection
  sargramostim : Given by injection
  tetanus peptide melanoma vaccine : Given by injection
- Arm III (12MP/6MHP): Patients receive 2 injections of multi-epitope peptide vaccine comprising multi-epitope melanoma peptide vaccine (12MP) and 6 melanoma helper peptides (6HP) emulsified with GM-CSF and ISA-51 (incomplete Freund's adjuvant) ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  multi-epitope melanoma peptide vaccine : Given by injection
  incomplete Freund's adjuvant : Given by injection
  sargramostim : Given by injection
  melanoma helper peptide vaccine : Given by injection
- Arm IV (6MHP): Patients receive 2 injections of multi-epitope peptide vaccine comprising melanoma helper peptide vaccine (6HP) emulsified with GM-CSF and ISA-51 (incomplete Freund's adjuvant) ID and SC on day 1 of weeks 1-3 and 1 injection at the primary site only on day 1 of weeks 5-7.
  incomplete Freund's adjuvant : Given by injection
  sargramostim : Given by injection
  melanoma helper peptide vaccine : Given by injection
Period: Overall Study
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Started | 47 | 43 | 37 | 48
Eligible | 43 | 36 | 33 | 42
Treated | 45 | 38 | 36 | 48
Eligible and Treated | 41 | 33 | 32 | 42
Have CTL Response Data | 40 | 30 | 29 | 41
Have Helper T Cell Response Data | 37 | 27 | 25 | 39
Completed | 1 | 2 | 0 | 3
Not Completed | 46 | 41 | 37 | 45
Not completed — Lack of Efficacy | 37 | 29 | 30 | 43
Not completed — Adverse Event | 4 | 4 | 3 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — No protocol therapy | 2 | 5 | 1 | 0
Not completed — others (not specified in the study) | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP) | Total
Number analyzed (Participants) | 41 | 33 | 32 | 42 | 148
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 86] | 69 [31 to 88] | 66 [32 to 89] | 64 [40 to 82] | 66 [31 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 11 | 17 | 60
  Male | 23 | 19 | 21 | 25 | 88
Region of Enrollment [Number; unit: participants]
  United States | 41 | 33 | 32 | 42 | 148

OUTCOME MEASURES:

1. Primary Outcome: Cytotoxic T-cell Lymphocytes (CTL) Response Rate
Description: Assessment of CTL response was based on a fold-increase in T cell response measure by interferon-gamma ELIspot assay.
Time Frame: Immune response was assessed at pre-registrtion, in weeks 1, 3, 5, 7, 8
Population: 140 eligible and treated patients who had CTL response data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Number analyzed (Participants) | 40 | 30 | 29 | 41
percentage of participants | 43 [27 to 59] | 47 [28 to 66] | 28 [13 to 47] | 5 [0.6 to 16.5]
Statistical Analysis 1: Comparison: Arm I (12MP) vs Arm II (12MP/Tet) vs Arm III (12MP/6MHP) vs Arm IV (6MHP); Compare CTL response rate among four arms. The null hypothesis is that CTL response is same in all four arms. Alternative hypothesis is that CTL response rate is different in at least one arm compared to other arms; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Helper T-cells Response to 6MHP
Description: Helper T cell response was evaluated by tritiated thymidine proliferation assay with fresh/cryopreserved PBL in the presence of each of the helper peptides.
Time Frame: Immune response was assessed at pre-registration, in weeks 1,3,5,7,8
Population: 128 eligible and treated patients who had data about helper T cell response were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Number analyzed (Participants) | 37 | 27 | 25 | 39
percentage of participants | 3 [0 to 14] | 0 [0 to 13] | 40 [21 to 61] | 41 [26 to 58]
Statistical Analysis 1: Comparison: Arm I (12MP) vs Arm II (12MP/Tet) vs Arm III (12MP/6MHP) vs Arm IV (6MHP); Compare HTL response rate to 6MHP among four arms. The null hypothesis is that HTL response is same in all four arms. Alternative hypothesis is that HTL response rate is different in at least one arm compared to other arms; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Helper T Cell Response to Tetanus
Description: as for outcome 2
Time Frame: Immune response was assessed at pre-registration, in weeks 1,3,5,7,8
Population: 128 eligible and treated patients who had data about HTL response to tetanus peptide were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Number analyzed (Participants) | 37 | 27 | 25 | 39
percentage of participants | 11 [3 to 25] | 59 [39 to 79] | 4 [0 to 20] | 0 [0 to 9]
Statistical Analysis 1: Comparison: Arm I (12MP) vs Arm II (12MP/Tet) vs Arm III (12MP/6MHP) vs Arm IV (6MHP); Compare HTL response rate to tetanus peptide among four arms. The null hypothesis is that HTL response is same in all four arms. Alternative hypothesis is that HTL response rate is different in at least one arm compared to other arms; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Objective Response Rate
Description: Tumor response was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Objective response rate is calculated as the number of patients with complete response (disappearance of all lesions) or partial response () divided by total number of evaluable patients.
Time Frame: Tumor response was assessed in weeks 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, and 6 months after last vaccination
Population: 148 eligible and treated patients were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Number analyzed (Participants) | 41 | 33 | 32 | 42
percentage of participants | 2.4 [0.06 to 12.8] | 3.0 [0.08 to 15.8] | 6.3 [0.8 to 20.8] | 7.1 [1.5 to 19.5]
Statistical Analysis 1: Comparison: Arm I (12MP) vs Arm II (12MP/Tet) vs Arm III (12MP/6MHP) vs Arm IV (6MHP); Compare objective response rate among four arms. The null hypothesis is that objective response rate is same in all four arms. Alternative hypothesis is that objective response rate is different in at least one arm compared to other arms; Test type: Superiority or Other; p = 0.741, Fisher Exact

5. Secondary Outcome: Median Overall Survival (OS)
Description: OS was defined as the time from registration to death from any cause.
Time Frame: assessed every 3 month within 2 years and every 6 months betwen 2 and 5 years
Population: 148 eligible and treated patients were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Number analyzed (Participants) | 41 | 33 | 32 | 42
months | 14.9 [10.1 to 18.6] | 10.2 [6.7 to 12.2] | 12.4 [4.8 to 16.8] | 11.1 [8.8 to 14.2]
Statistical Analysis 1: Comparison: Arm I (12MP) vs Arm II (12MP/Tet) vs Arm III (12MP/6MHP) vs Arm IV (6MHP); Compare overall survival curves among four arms; Test type: Superiority or Other; p = 0.532, Log Rank

ADVERSE EVENTS:
Time Frame: Assessed at the end of each cycle while on treatment and at 30 days following the last dose of treatment. Reported every 3 months within 2 years of study entry, and every 6 months between 2-5 years of study entry
Description: All patients who received protocol therapy were evaluated for toxicity, regardless of eligibility.
Arm/Group | Arm I (12MP) | Arm II (12MP/Tet) | Arm III (12MP/6MHP) | Arm IV (6MHP)
Serious Adverse Events (participants affected / at risk) | 6/45 | 9/38 | 6/36 | 4/48
Other Adverse Events (participants affected / at risk) | 36/45 | 28/38 | 28/36 | 33/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (12MP) (N=45) | Arm II (12MP/Tet) (N=38) | Arm III (12MP/6MHP) (N=36) | Arm IV (6MHP) (N=48)
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Leukocytes decreased) (Investigations) | 1 | 1 | 0 | 0
Lymphopenia (Investigations) | 1 | 1 | 1 | 0
Neutropenia (Neutrophils decreased) (Investigations) | 1 | 0 | 0 | 0
Cardiac troponin I (cTnI) (Investigations) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 4 | 5 | 1
Injection site reaction (General disorders) | 2 | 3 | 0 | 2
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 1 | 0 | 0 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase (ALT, SGPT) (Investigations) | 0 | 0 | 2 | 0
Aspartate aminotransferase (AST, SGOT) (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic/Laboratory-other (Investigations) | 0 | 0 | 1 | 0
Central nervous system (CNS) cerebrovascular ischemia (Nervous system disorders) | 0 | 1 | 0 | 0
Abdomen, pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Head/headache (Nervous system disorders) | 0 | 1 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (12MP) (N=45) | Arm II (12MP/Tet) (N=38) | Arm III (12MP/6MHP) (N=36) | Arm IV (6MHP) (N=48)
Leukopenia (Leukocytes decreased) (Investigations) | 3 | 5 | 1 | 0
Lymphopenia (Investigations) | 2 | 8 | 6 | 4
Neutropenia (Neutrophils decreased) (Investigations) | 0 | 2 | 0 | 1
Thrombocytopenia (Platelets decreased) (Investigations) | 2 | 3 | 2 | 1
Fatigue (General disorders) | 9 | 11 | 10 | 7
Fever w/o neutropenia (General disorders) | 1 | 4 | 2 | 0
Rigors/chills (General disorders) | 1 | 5 | 4 | 2
Sweating (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1
Injection site reaction (General disorders) | 28 | 20 | 18 | 18
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 2 | 5 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 6 | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Alkaline phosphatase increased (Investigations) | 4 | 3 | 2 | 4
Aspartate aminotransferase increased (AST, SGOT) (Investigations) | 3 | 5 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 2 | 2 | 0
Creatinine increased (Investigations) | 2 | 3 | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Metabolic/Laboratory-other (Investigations) | 2 | 2 | 5 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0
Head/headache (Nervous system disorders) | 5 | 5 | 3 | 2
Joint, pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Alanine aminotransferase increased (ALT, SGPT) (Investigations) | 2 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No